CLINICAL TRIAL: NCT02436694
Title: Can the Association of Dexamethasone and Local Anaesthetic in a Single-shot Femoral and Sciatic Nerve Block Improve Analgesia Postoperatively in Patients Submitted to Total Knee Arthroplasty
Brief Title: Nerve Blocks With Dexamethasone and Local Anaesthetic to Improve Postoperative Analgesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Hospitalar do Porto (Other)
Responsible Party: Principal Investigator, Marta Carvalho, MD, Centro Hospitalar do Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014.236(174-DEFI/199-CES)
Record Dates: First submitted 2015-04-01; First posted 2015-05-07 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Nerve Block
Keywords: Dexamethasone; Perineural
MeSH Terms: interventions — Nerve Block; Anesthetics, Local; Dexamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local Anesthetic ropivacaíne (Active Comparator): Femoral nerve block with ropivacaine 0.375% and sciatic nerve block with ropivacaine 0.2%
  Interventions: Drug: Local Anesthetic ropivacaíne
- Perineural Dexamethasone (Experimental): Femoral nerve block with ropivacaine 0.375% and perineural dexamethasone and sciatic nerve block with ropivacaine 0.2% and perineural dexamethasone
  Interventions: Drug: Local Anesthetic ropivacaíne; Drug: Perineural Dexamethasone

INTERVENTIONS:
Drug: Local Anesthetic ropivacaíne — Femoral and sciatic nerve block with ropivacaíne
  Other Names: Nerve block with local anesthetic
Drug: Perineural Dexamethasone — Addition of perineural dexamethasone to local anesthetic for femoral and sciatic nerve block
  Other Names: Nerve block with local anesthetic and dexamethasone
  Arms: Perineural Dexamethasone

SUMMARY:
Can the association of dexamethasone to the local anaesthetic in a single-shot femoral and sciatic nerve block improve analgesia postoperatively in patients submitted to total knee arthroplasty? Primary aim: Evaluate the efficacy of the association of dexamethasone to the local anaesthetic in a SSFNB and SSSNB in reducing pain scores, assessed by VAS.

Outcome measures: Mean pain scores in both groups. Secondary aims: Evaluate opioid consumption in the postoperative period (8- 12h, 24h, 48h) and assess incidence of side effects and complications (numbness, paraesthesias, weakness, site infection, haematoma and falls).

DETAILED DESCRIPTION:
All blocks are performed using nerve stimulation technique. For the SSFNB, the paravascular approach will be used to identify the femoral nerve.15 A positive location is considered when quadriceps contraction (patellar elevation) is elicited with a current of 0.4 mA or less, and 30mL of ropivacaine 0.375%, with or without 4mg of dexamethasone are injected, according to the randomization.

For the SSSNB the anterior approach will be chosen.16 The common peroneal or the tibial nerves are identified, respectively by dorsiflexion or plantar flexion of the foot, with a current of 0.4 mA or less. Depending on the allocated group, 20mL of ropivacaine 0.2%, with or without 4mg of dexamethasone are then injected. Blocks success should be assessed by the absence of thermal sensitivity on the anterior region of the thigh and the dorsum of the foot 10 minutes after the block.

The participating anaesthesiologists may use the ultrasound for visual guidance but should also use the nerve stimulator in order to maintain the homogeneity of the procedure.

Patients will then have an intravenous induction to general anesthesia, being the maintenance assured with either Desflurane or Sevoflurane. Thirty minutes before the end of the procedure all patients are given paracetamol 1000mg and ketorolac 30mg. Total doses of intraoperative analgesics are recorded.

Before surgery all patients will be explained how to use the PCA, which is connected after arrival to the post-anesthesia unit (PACU). The PCA is programmed for 1mg bolus as required by the patient, with a lockout period of 7 minutes. In what concerns the remaining post-operative analgesia, both groups are prescribed paracetamol 1000mg q8h, diclofenac 50mg q12h, and as rescue strategy, tramadol 100mg q6h.

The demographic data as well as the information of the anesthetic form is recorded in an excel table. After surgery, at 8-12h, 24h and 48h (+/-2h) pain is evaluated using a standard 100mm VAS. Consumption of morphine and other rescue analgesia is recorded in the same time periods, as well as the complications and side-effects previously determined.

The primary outcome is pain assessed by VAS (1-100mm - continuous variable), measured ate 8-12h, 24h and 48h. Difference in mean values for both groups will be measured. Morphine consumption is measured in milligrams, and the mean consumption of both groups is analysed. Side-effects and complications will be reported and their incidence calculated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted foi unilaterla total knee arthroplasty

Exclusion Criteria:

* Refusal/Incapacity to give informed consent
* Contra-indication to general anesthesia
* Infection at needle insertion site
* Coagulation disorders
* Pre-existing neurologic disorders
* Known allergy to any of the drugs from the protocol
* ASA status >3
* Weight<50kg
* BMI>40
* Inability to understand or use VAS pain score

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Quantification of Pain by VAS | 48 hours
  Pain assessed by VAS

SECONDARY OUTCOMES:
Morphine consumption in mg | 48 hours
  Morphine consumption in PCA measured in mg
Side-effects (numbness, paraesthesias, weakness, site infection, haematoma and falls) | 48 hours
Complications from technique (Motor ou sensitive changes, infection, nausea) | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Raul carvalho, MD, Study Director — Centro Hospitalar do Porto
Locations (1):
- Centro Hospitalar do Porto, Porto, Porto District, Portugal